CLINICAL TRIAL: NCT00311961
Title: A Comparison of Intravenous Versus Oral Administration of Prednisolone in the Treatment of Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Intravenous Versus Oral Administration of Prednisolone in Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isala (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IK-001
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Exacerbations; Corticosteroids; Oral; Intravenous; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Prednisolone

INTERVENTIONS:
Drug: Intravenous prednisolone
Drug: Oral prednisolone

SUMMARY:
Treatment with systemic corticosteroids for acute exacerbations of COPD results in the improvement of clinical outcomes. The optimal route of administration has not been rigorously studied in COPD. Upon hospitalization, corticosteroids are administered intravenously in many hospitals. Oral administration is more convenient, though, because there is no need for intravenous access, less personnel is required for starting and monitoring therapy, and material costs are smaller.

The investigators hypothesized that oral administration is not inferior to intravenous administration of prednisolone in the treatment of patients hospitalized for an acute exacerbation of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Exacerbation of COPD (at least Global Initiative for Chronic Obstructive Lung Disease [GOLD] severity stage II)
* Smoking history of > 10 pack years

Exclusion Criteria:

* Signs of severe exacerbation (arterial pH < 7.26 or pCO2 > 9.3 kPa)
* History of asthma
* Significant or unstable co-morbidity
* Participated in another study 4 weeks before admission
* Previously randomized to this study
* Findings on chest radiography other than those fitting with signs of COPD
* Known hypersensitivity to prednisolone
* Non-compliant

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 256
Dates: Start 2001-06; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Treatment failure defined as: death from any cause
admission to the intensive care unit
readmission to the hospital because of COPD
and the necessity to intensify pharmacologic treatment

SECONDARY OUTCOMES:
Changes in forced expiratory volume in 1 second (FEV1)
St. George's Respiratory Questionnaire (SGRQ) scores
Clinical COPD Questionnaire (CCQ) scores
and length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jan WK van den Berg, MD, PhD, Principal Investigator — Isala; Ynze P de Jong, MD, Principal Investigator — Isala
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Derived] de Jong YP, Uil SM, Grotjohan HP, Postma DS, Kerstjens HA, van den Berg JW. Oral or IV prednisolone in the treatment of COPD exacerbations: a randomized, controlled, double-blind study. Chest. 2007 Dec;132(6):1741-7. doi: 10.1378/chest.07-0208. Epub 2007 Jul 23. PMID 17646228